CLINICAL TRIAL: NCT06088732
Title: Effects of Acute Exercise and Ibuprofen on Symptoms, Immunity, and Neural Circuits in Bipolar Depression
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2023-001
Record Dates: First submitted 2023-10-12; First posted 2023-10-18 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder | interventions — Ibuprofen; RE1-silencing transcription factor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Session 1 (Experimental): Exercise (30 min on bicycle ergometer at 60% peak power output) and a single oral dose 800mg of ibuprofen
  Interventions: Other: Exercise Session; Drug: Ibuprofen 800 mg
- Session 2 (Active Comparator): Exercise (30 min on bicycle ergometer at 60% peak power output) and matching placebo
  Interventions: Other: Exercise Session; Drug: Placebo
- Session 3 (Active Comparator): 30 minutes rest (sitting in chair) and a single oral dose 800mg of ibuprofen
  Interventions: Drug: Ibuprofen 800 mg; Other: Rest
- Session 4 (Placebo Comparator): 30 minutes rest (sitting in chair) and matching placebo
  Interventions: Other: Rest; Drug: Placebo

INTERVENTIONS:
Other: Exercise Session — 30 min cycling on bicycle ergometer at 60% peak power output
  Arms: Session 1; Session 2
Drug: Ibuprofen 800 mg — A single oral dose of Ibuprofen
  Arms: Session 1; Session 3
Other: Rest — Resting for 30 min in chair
  Arms: Session 3; Session 4
Drug: Placebo — Matched placebo
  Arms: Session 2; Session 4

SUMMARY:
This is a 2x2, within-subjects, cross-over trial to test the anti-depressant effects of acute exercise in 20 participants with bipolar depression. Participants will complete four experimental sessions, two with an exercise challenge and two with a resting control condition in a counterbalanced order. Participants will receive either 800mg of ibuprofen or placebo before exercise or rest in order to test whether blocking the inflammatory response to exercise interferes with the neural and psychological effects of exercise.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Has an established residence and phone
3. Agrees to and is eligible for behavioral testing, magnetic resonance imaging, and blood draws.
4. Stated willingness to comply with all study procedures and lifestyle considerations (see Section 5.3, Lifestyle Considerations) and availability for the duration of the study
5. Males and females; Age 18-55 years
6. DSM-V diagnosis of bipolar disorder
7. Has a current major depressive episode
8. Depression at enrollment of sufficient severity to score > 11 on the QIDS
9. Be stably medicated for at least 4 weeks (a non-medicated subject may be included in the study if judged to be appropriate in the medical/psychiatric opinion of the investigator)
10. BMI between 18.5 and 35

Exclusion Criteria:

1. Diagnosis of any other major psychiatric disorder such as schizoaffective disorder, schizophrenia, or current psychotic depression
2. A history of bipolar disorder with rapid cycling
3. Concurrent manic symptoms of sufficient severity to pose a substantial risk of the development of a manic episode (>19 on the YMRS)
4. Current drug or alcohol or substance use disorder moderate or severe, except nicotine (within 6 months for severe use disorder; 2 months for moderate use disorder)
5. Volunteers currently receiving more than 4 mood-relevant psychotropic medications in a daily regimen (since this may signify a more brittle or complex clinical state)
6. Taking any of the following medications: medications with significant interactions with ibuprofen; immune-modulating medications (e.g. oral steroids); regular use of NSAIDs (> 3 times per week)
7. Current or prior cardiac disease, cardiac arrhythmia (e.g. supraventricular tachycardia, atrial fibrillation, ventricular fibrillation), or history of cardiac ablation therapy
8. Unstable medical condition, including significant respiratory disease (e.g., asthma, reactive airway disease (i.e., exercise induced asthma), or chronic obstructive pulmonary disease (COPD)), liver disease, hypothyroidism (i.e., condition not adequately stabilized for 3 months), or other conditions likely to require hospitalization or with a life expectancy of < 6 months (e.g., cancer).
9. History of claustrophobia that would prevent participation in imaging scans
10. Actively suicidal, as defined by expressive ideation with a plan and intent for suicide or developing suicidal ideation that requires immediate medical or treatment intervention or a suicide attempt within the previous six months
11. Participants who endorse a history of moderate to severe traumatic brain injury (>30 min. loss of consciousness or >24 hours posttraumatic amnesia) or other neurocognitive disorder with evidence of neurological deficits
12. Inadequate understanding of English
13. Currently pregnant or breast-feeding; fecund women not using adequate contraceptive methods; plan to become pregnant within 12 months
14. Metal in the body (e.g. history of working as a sheet metal worker) or pacemaker which is a contra-indication to magnetic resonance imaging
15. Has epilepsy, a neuromuscular disorder, or tardive dyskinesia
16. Has a chronic infectious illness
17. Requires immediate hospitalization for psychiatric disorder
18. Requires medications for a general medical condition that contraindicate any study medication
19. Receiving or have received during the index episode vagus nerve stimulation, electroconvulsive therapy, transcranial magnetic stimulation, or other somatic treatments
20. Allergy to, or other medical contraindication to ibuprofen (e.g. stomach ulcers)
21. Symptoms of myalgic encephalomyelitis/chronic fatigue syndrome or "long-COVID".
22. Current use of medications or dietary supplements for weight or appetite control, whether prescribed or not
23. Ulcerative colitis, Crohn's disease or other autoimmune disorder (except treated hypothyroidism)
24. Activity restrictions that limit the subject's ability to engage in intense physical activity
25. Use of beta-blockers, calcium channel inhibitors, or other heart-modulating medications (e.g., amiodarone)
26. Clinically significant abnormality on EKG
27. Hypertension, hepatitis, renal dysfunction, and/or anemia of sufficient severity to pose a risk to the participant
28. Moderate or heavy smoker based on Fagerstrom
29. Resting heart rate >100 beats per minute, systolic blood pressure > 160 mmHg, diastolic blood pressure > 100 mmHg
30. Clinically significant screening laboratory abnormalities not covered above
31. Any reason not listed herein that would make participation in the study hazardous

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Inflammation | Difference between IL-6 at baseline and two hours post intervention
  Serum concentrations of interleukin 6 (IL-6)
Neural Response to Reward Anticipation | One hour post intervention
  Percent Signal Change in Ventral Striatum During Monetary Incentive Delay

SECONDARY OUTCOMES:
Neural Response to Reward Receipt | One hour post intervention
  Percent Signal Change in Ventral Striatum During Monetary Incentive Delay (MID) task
Brain Volume | One hour post intervention
  Gray Matter Volume of the Hippocampus
Inflammation | Difference between TNF at baseline and two hours post intervention
  Serum concentrations of tumor necrosis factor (TNF)
Inflammation | Difference between IL-10 at baseline and two hours post intervention
  Serum concentrations of interleukin 10 (IL-10)
Anhedonia | Difference between SHAPS scores at baseline and two hours post intervention
  Score on the Snaith-Hamilton Pleasure Scale (SHAPS). Higher scores indicate greater anhedonia. Score range from 0-14.

CONTACTS AND LOCATIONS:
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided